CLINICAL TRIAL: NCT04500912
Title: Comparison of the Supraflex Cruz 60 Micron Stent Strut Versus the Ultimaster Tansei 80 Micron Stent Strut in High Bleeding Risk PCI Population
Brief Title: Comparison of the Supraflex Cruz 60 Micron Versus the Ultimaster Tansei 80 Micron in HBR PCI Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pieter C.Smits (Other)
Collaborators: Sahajanand Medical Technologies Limited (Industry)
Responsible Party: Sponsor-Investigator, Pieter C.Smits, MD, PhD, Research Maatschap Cardiologen Rotterdam Zuid
Organization: Research Maatschap Cardiologen Rotterdam Zuid (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL73419.100.20
Record Dates: First submitted 2020-07-26; First posted 2020-08-05 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Cardiac Disease; PCI; High Bleeding Risk
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patient will be blinded for the stent that is used
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supraflex Cruz stent (Active Comparator): Randomization to Supraflex Cruz stent
  Interventions: Device: Supraflex Cruz 60 Micron
- Ultimaster Tansei stent (Active Comparator): Randomization to Ultimaster Tansei stent
  Interventions: Device: Ultimaster Tansei 80 Micron

INTERVENTIONS:
Device: Supraflex Cruz 60 Micron — percutaneous coronary intervention
  Arms: Supraflex Cruz stent
Device: Ultimaster Tansei 80 Micron — percutaneous coronary intervention
  Arms: Ultimaster Tansei stent

SUMMARY:
The study compares the outcome of the ultrathin stent strut Supraflex Cruz stent to the thin stent strut Ultimaster Tansei stent in a PCI population at high risk for bleeding (HBR).

DETAILED DESCRIPTION:
Study design: An Investigator-initiated, multi-center, randomized clinical trial in HBR patients receiving PCI with Supraflex Cruz or Ultimaster Tansei stents

Study population: 2 x 368 (736) patients, who undergo a PCI and are at high risk for bleeding (HBR).

Intervention: Patients are treated according to the randomized regimen at index PCI and at planned staged procedures. Either with the ultrathin stent strut Supraflex Cruz stent to the thin stent strut Ultimaster Tansei stent

DAPT treatment (combination and duration) is according to the Guidelines of the European Society of Cardiology for Myocardial Revascularization.

Follow-up is scheduled at 1 month, 6 months and 12 months post index PCI procedure.

Primary study parameters/outcome of the study:

The primary endpoint Net Adverse Clinical Endpoints (NACE) defined as a composite of cardiovascular death, myocardial infarction, target vessel revascularization, stroke and bleeding events defined as BARC 3 or 5 at 12 months follow-up after the index PCI.

ELIGIBILITY:
Inclusion criteria:

Patients are eligible for inclusion into the study if the following criteria are met.

* Patients of 18 years and above
* Written or witnessed oral consent to participate in the study
* Native coronary artery lesions eligible for PCI with stents with no restrictions in number of lesions and stents, vessel size or lesion complexity, apart from stent thrombosis.
* Patients at high risk for bleeding according to the HBR ARC criteria: Patients meet the HBR ARC criteria if ≥1 major or ≥2 minor criteria are met.

Major HBR criteria are the following:

* Clinical indication for treatment with oral anticoagulants (OAC/NOAC) for at least 12 months
* Severe or end-stage chronic kidney failure (GFR ≤ 30 ml/min)
* Hemoglobin (Hb) level at screening < 11g/dl or < 6.8 mmol/l
* Spontaneous bleeding requiring hospitalization or transfusion in the past 6 months or at any time, if recurrent
* Moderate or severe baseline true thrombocytopenia (platelet count <100 *10^9/L)
* History of chronic bleeding diathesis, like: leukemia, haemophilia, vitamin K deficiency, Factor V or VII deficiency etc.
* Liver cirrhosis with portal hypertension
* Active malignancy (other than skin) within the past 12 months
* Spontaneous intracranial haemorrhage ICH (at any time)
* Traumatic intracranial haemorrhage ICH within 12 months
* Presence of a brain arterio-venous malformation (AVM)
* Moderate or severe ischemic stroke within the past 6 months
* Nondeferrable major surgery on DAPT after PCI
* Recent major surgery or major trauma within 30 d before PCI

Minor HBR criteria are the following:

* Age ≥ 75 years
* Moderate chronic kidney disease (GFR >30 and <60 ml/min)
* Hemoglobin (Hb) 11-12.9 g/dL / 6.8-8.0 mmol/l for men and 11-11.9 g/dL / 6.8-7.4 mmol/l for women
* Any ischemic stroke at any time not meeting the major criterion
* Spontaneous bleeding requiring hospitalization or transfusion within the past 12 months
* Need for chronic treatment with steroids or non-steroidal anti-inflammatory drugs

Exclusion criteria:

Patients are not eligible if any of the following applies:

* Treated with stents other than Supraflex Cruz or Ultimaster within 6 months prior to index procedure
* Treatment of lesions with stent thrombosis
* Treatment of venous or arterial coronary grafts
* Treated for stent thrombosis in 12 months prior to index PCI procedure
* Treated with a bioresorbable scaffold 3 years before index PCI procedure
* Cardiogenic shock at index procedure
* Active SARS-CoV-2 infection or suspicion of SARS-CoV-2 infection
* Cannot provide written informed consent
* Under judicial protection, tutorship or curatorship
* Unable to understand and follow study-related instructions or unable to comply with study protocol
* Active bleeding requiring medical attention (BARC≥2) at index PCI
* Life expectancy less than one year
* Known hypersensitivity or allergy for aspirin, clopidogrel, ticagrelor, prasugrel, cobalt chromium or sirolimus
* Any anticipated PCI after index PCI, unless planned and scheduled at index PCI
* Participation in another stent or drug trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 736 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Net Adverse Clinical Endpoints (NACE) | 1 year
  The primary endpoint Net Adverse Clinical Endpoints (NACE) defined as a composite of cardiovascular death, myocardial infarction, target vessel revascularization, stroke and bleeding events defined as BARC 3 or 5 at 12 months follow-up after the index PCI.

SECONDARY OUTCOMES:
Major adverse cardiac and cerebral events (MACCE) | 1 year
  Major adverse cardiac and cerebral events (MACCE) defined as a composite of cardiac death, myocardial infarction, target vessel revascularization and stroke
Major or clinically relevant non-major bleeding (MCB) | 1 year
  Major or clinically relevant non-major bleeding (MCB) defined as a composite of type 2, 3 and 5 BARC bleeding events
Target Lesion Failure (TLF) | 1 year
  Target Lesion Failure (TLF) is defined as cardiac death, myocardial infarction attributed to the target vessel and clinically indicated target lesion revascularization
Target vessel failure (TVF) | 1 year
  Target Vessel Failure (TVF) is defined as cardiac death, myocardial infarction attributed to the target vessel and clinically indicated target vessel revascularization
The composite of cardiovascular death, myocardial infarction and stroke | 1 year
  The composite endpoint of cardiovascular death, myocardial infarction and stroke
The composite of cardiovascular death, myocardial infarction, stroke and major bleed BARC 3 and 5 | 1 year
  The composite of cardiovascular death, myocardial infarction, stroke and major bleed according to BARC 3 and 5
Stent thrombosis | 1 year
  Stent thrombosis according to the ARC definitions
Myocardial infarction | 1 year
  Myocardial infarction.
Urgent target vessel revascularization | 1 year
  Urgent target vessel revascularization.
Non-target vessel revascularization | 1 year
  Non-target vessel revascularization.
Clinically indicated target vessel revascularization | 1 year
  Clinically indicated target vessel revascularization.
Bleeding events | 1 year
  Bleeding events according to the BARC, TIMI and GUSTO classification
Transfusion rates | 1 year
  Transfusion rates both in patients with and/or without clinically detected over bleeding
Event rates according to the PRECISE-DAPT | 1 year
  Event rates according to the PRECISE-DAPT score
Procedural success | At completion of the baseline PCI
  Procedural success is defined as angiographic success with no in-hospital MACE, defined as death, MI with new Q-waves on electrocardiogram (ECG) or urgent target vessel revascularization (TVR) (including both repeat PCI and coronary artery bypass graft surgery (CABG)
Device success | At discharge of baseline hospitalisation, on average 3 days
  Device success (applying a lesion-level analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Smits, MD, PhD, Principal Investigator — Research Maatschap Cardiologen Rotterdam Zuid
Locations (11):
- Netherlands (11):
  - Jeroen Bosch ziekenhuis, 's-Hertogenbosch
  - Meander ziekenhuis, Amersfoort
  - Rijnstate ziekenhuis, Arnhem
  - Tergooi ziekenhuis Blaricum, Blaricum
  - Amphia Ziekenhuis, Breda
  - Albert Schweitzer ziekenhuis, Dordrecht
  - Catherina ziekenhuis, Eindhoven
  - MCL Leeuwarden, Leeuwarden
  - St.Antonius ziekenhuis, Nieuwegein
  - Maasstadziekenhuis, Rotterdam
  - Ziekenhuis Zorgsaam, Terneuzen

REFERENCES:
- [Derived] Smits PC, Tonino PAL, Hofma SH, van Kuijk JP, Spano F, Al Mafragi A, Pisters R, Polad J, Bogaerts K, Oemrawsingh RM, Paradies V. Comparison of Ultrathin- Versus Thin-Strut Stents in Patients With High Bleeding Risk PCI: Results From the COMPARE 60/80 HBR Trial: An Open-Label, Randomized, Controlled Trial. Circ Cardiovasc Interv. 2024 Oct;17(10):e014042. doi: 10.1161/CIRCINTERVENTIONS.123.014042. Epub 2024 Oct 1. PMID 39351676
- [Derived] Capodanno D. Another Coronary Stent for Patients at High Bleeding Risk. JACC Cardiovasc Interv. 2021 Sep 13;14(17):1884-1887. doi: 10.1016/j.jcin.2021.07.028. No abstract available. PMID 34503738